CLINICAL TRIAL: NCT01147120
Title: CAM Referral and Outcomes: Chronic Low Back Pain in Urban and Rural Primary Care
Brief Title: Chronic Low Back Pain and Primary Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William G Elder JR (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, William G Elder JR, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21AT004544-01A2 (NIH); 1R21AT004544-01A2 (NIH)
Record Dates: First submitted 2010-03-30; First posted 2010-06-22 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progressive Muscle Relaxation (Active Comparator)
  Interventions: Behavioral: Progressive Muscle Relaxation (PMR)
- Clinical Massage Therapy (Active Comparator)
  Interventions: Procedure: Clinical Massage Therapy (CMT)

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation (PMR) — Progressive Muscle Relaxation (PMR) will be recorded on PDAs integrated with EMA software and offered to patients who will be instructed in the techniques and PDA use by study coordinators. They will be instructed to practice 25 minutes/day the first two weeks, 35 minutes/day weeks 3 and 4, and 45 minutes/day weeks 5 through 12. These time periods (25/35/45 minute) were selected to allow a more gradual acclimation to PMR.
  Arms: Progressive Muscle Relaxation
Procedure: Clinical Massage Therapy (CMT) — PCPs will have the opportunity to refer patients with CLBP to local Licensed Massage Therapists (LMTs) to receive up to 10 clinical massage sessions over a 12-week period. CMT will be provided at no cost to the patients. At their first two sessions, the LMT will evaluate the patient and, with the patient, estimate the number of sessions and determine treatment goals. Based on previous literature, 10 sessions are anticipated over an average 12-week period. However, treatment will vary depending on assessment and progress. At the end of the treatment period, the patients will receive a list of all participating LMTs to facilitate patients' continued or future participation in massage therapy.
  Arms: Clinical Massage Therapy

SUMMARY:
Kentucky ranks 2nd in disability among states, with chronic low back pain (CLBP) as a major disability, especially in the investigators rural areas. Kentucky and U.S. health care providers need alternative and effective treatments. Following NCCAM strategic research recommendations, this study will investigate health services outcomes of complementary and alternative medicine (CAM) therapies in an existing primary care practice-based research network (PBRN). The Patients with CLBP are often willing to try therapeutic options outside the conventional medical spectrum. Massage and relaxation therapies have demonstrated fairly good efficacy in controlled trials but their effectiveness in the "real world" of primary care is only beginning to be evaluated. The long-term goal of the proposed project builds on the foundation of these two established therapies to improve treatment of chronic low back pain (CLBP) in primary care practices. Two alternative (CAM) therapies, progressive muscle relaxation (PMR) and clinical massage therapy (CMT), will be studied. The short-term objectives of the proposed project are to: (1) examine outcomes of CAM for patients with CLBP referred from primary care practices, and (2) better understand physician decision-making to recommend CAM therapy for CLBP. Specific Aim 1 will evaluate improvement in health-related outcomes for patients with CLBP when referred to PMR or CMT from primary care. Specific Aim 2 will explore selected factors in primary care physicians' decisions to recommend CAM therapy to these patients. The proposed study is unique in that it addresses "real life" clinical situations and decision-making in both urban and rural clinical practices within an existing PBRN. Should such CAM referral prove successful for ameliorating CLBP, it would provide relatively low cost, non-addictive treatment options for inclusion in the repertoire of primary care physicians.

DETAILED DESCRIPTION:
The proposed study will investigate health related outcomes of two CAM treatments recommended by primary care physicians for CLBP, and explore selected elements in the decision process to recommend or not recommend one of two CAM treatments.

Patients and primary care physicians (PCPs) will participate from metropolitan and nonmetropolitan central Kentucky practices of the Kentucky Ambulatory Network (KAN), Kentucky's statewide primary care practice-based research network (PBRN). Each practice will have a patient participant enrollment period of four weeks. Patients with CLBP who have a visit during the enrollment period in a practice may be eligible to participate in the study, and participating PCPs will be invited to recommend as many eligible patients as they feel comfortable. During patient visits, the PCP may offer a recommendation to the patient to receive PMR or CMT. Patients who agree will be recruited by the KAN/CAM project team staff. Patients who enroll in the CAM recommendation study will receive a 12-week course of PMR or CMT treatments. Outcomes will be measured at three time points: baseline, 12 weeks, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a visit with the physician during the 4-week study referral period for that practice
* Be 21 years of age or older on the date of the visit
* According to the physician, currently have CLBP
* Have been a patient in the practice for at least 3 months
* Have a life expectancy of 6 months or more

Exclusion Criteria:

* Not have a current or past history of psychosis
* Not be pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2009-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline, 12 Weeks, and 24 Weeks
  Survey completed at Baseline, 12 Weeks, and 24 Weeks
Short Form 36 (SF-36) | Baseline, 12 Weeks, and 24 Weeks
  Health related quality of life survey
Faces Pain Scale - Revised (FPS-R) | Baseline, 12 Weeks, and 24 Weeks
  Survey

SECONDARY OUTCOMES:
Pain Medication Questionnaire (PMQ) - subset | Baseline, 12 Weeks, and 24 Weeks
  Survey
Expectations for and Satisfaction with Therapies | Baseline and 12 Weeks
  Survey
Tampa Scale of Kinesiophobia (TSK) - Subset | Baseline, 12 Weeks, and 24 Weeks
  Survey
Patient Perceptions of CAM Therapy | Baseline, 12 Weeks, and 24 Weeks
  Survey
Physician Perceptions of CAM Therapy | Baseline
  Survey
Physician Point-of-Care Card | 4 weeks per practice (Identify and screen for possible patients)
  CLBP visit description and reasons to recommend patients for this therapy study.

CONTACTS AND LOCATIONS:
Overall Officials: William G Elder, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Department of Family and Community Medicine; University of Kentucky, Lexington, Kentucky, United States